CLINICAL TRIAL: NCT05177835
Title: A Follow-up Phase II Open-label Study to Evaluate the Long-term Safety and Efficacy Profile of ABX464 Given at 25 mg Once Daily in Subjects With Moderate to Severe Active Ulcerative Colitis
Brief Title: Long-term Safety and Efficacy Profile of ABX464 in Subjects With Moderate to Severe Active Ulcerative Colitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABX464-108
Record Dates: First submitted 2021-12-15; First posted 2022-01-05 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis
Keywords: Moderate to severe ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ABX464

STUDY DESIGN:
Intervention Model Description: Open Label Follow-up Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABX464 -25mg (Experimental): All subjects will receive ABX464 given at 25 mg QD.
  Interventions: Drug: ABX464

INTERVENTIONS:
Drug: ABX464 — All subjects will receive ABX464 given at 25 mg QD.

SUMMARY:
This study is an open-label study aiming at evaluating the long-term safety and the efficacy profile of ABX464 given once a day (QD) at 25 mg in subjects who have been previously enrolled in the ABX464-102 or ABX464-104 studies (OLE and maintenance studies) and who are willing to continue their treatment.

All subjects will receive ABX464 given at 25 mg QD. The enrolment in this long-term study will be based on the endoscopic improvement, the willingness of the subject to carry on his/her participation and also based on investigator's judgement.

Subjects will be treated with ABX464 for a maximum period of 54 months. Subjects will be followed up quarterly. After the treatment period, subjects will be followed for 4 additional weeks for safety purposes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who previously completed the ABX464-102 or ABX464-104 clinical studies
* Subjects should be in endoscopic improvement with a rectal bleeding sub-score = 0 point at the end of treatment period in the previous study (ABX464-102 or ABX464-104). Endoscopic improvement is defined as: a Mayo endoscopic sub score of ≤1 ;
* Subjects able and willing to comply with study visits and procedures;
* Subjects must understand, sign and date the written voluntary informed consent form at the visit prior to any protocol-specific procedures;
* 5. Women of childbearing potential and men receiving the study treatment and their partners must agree to continue a highly effective contraceptive method during the study and for 6 months (180 days) after end of study or early termination. Women must be surgically sterile or if of childbearing potential must use a highly effective contraceptive method. Women of childbearing potential (WOCBP) will enter the study after confirmed menstrual period and a negative pregnancy test. Highly effective methods of contraception include true abstinence, intrauterine device (IUD) or hormonal contraception aiming at inhibition of ovulation, intrauterine hormone releasing system, bilateral tubal ligation, vasectomized partner. True abstinence is defined when this is in line with the preferred and usual lifestyle of the subject. In each case of delayed menstrual period (over one month between menstruations) confirmation of absence of pregnancy is required. This recommendation also applies to WOCBP with infrequent or irregular menstrual cycle. Female and male subjects must not be planning pregnancy during the trial and for 6 months post completion of their participation in the trial. In addition, male subjects should use condom during the trial and for 6 months (180 days) post completion of their participation in the study. Male subjects must not donate sperm as long as contraception is required. For the purpose of this protocol, a woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. Finally, a man is considered fertile after puberty unless permanently sterile by bilateral orchidectomy;
* Subjects should be affiliated to a social security regimen (for French sites only).

Exclusion Criteria:

* Subjects who have developed any major illness/condition or evidence of an unstable clinical condition (except UC) that, in the investigator's judgment, will substantially increase the risk to the participant if he or she participates in the study
* Subjects with any other severe acute or chronic medical or psychiatric condition or laboratory or electrocardiogram (ECG) abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study
* Subjects who are participating or plan to participate in other investigational studies (other than induction study) during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events in ABX464 treated subjects | From Baseline to a maximum period of 54 months
  To evaluate the long-term safety of ABX464 given at 25 mg once daily in subjects with Moderate to Severe Active Ulcerative Colitis.

SECONDARY OUTCOMES:
Percentage of subjects reaching clinical remission at yearly visits. | From Baseline to a maximum period of 54 months
  To evaluate the long-term effect of ABX464 on clinical remission
Percentage of subjects reaching endoscopic remission at yearly visits | From Baseline to a maximum period of 54 months
  To evaluate the long-term effect of ABX464 on endoscopic remission
Percentage of subjects reaching clinical response at yearly visits | From Baseline to a maximum period of 54 months
  To evaluate the long-term effect of ABX464 on clinical response
Percentage of subjects reaching endoscopic improvement at yearly visits | From Baseline to a maximum period of 54 months
  To evaluate the long-term effect of ABX464 on endoscopic improvement

CONTACTS AND LOCATIONS:
Overall Officials: Bram Verstockt, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (46):
- Austria (2):
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Medical University of Vienna, Vienna
- Belgium (2):
  - Antwerp University Hospital, Antwerp
  - UZ Leuven, Leuven
- South Edmonton Gastroenterology, Edmonton, Canada
- Czechia (2):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Nemocnice Slany, Slaný
- France (5):
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - Centre Hospitalier Universitaire De Montpellier, Montpellier
  - CHU Nantes - Hôtel Dieu, Nantes
  - Institut des MICI, Neuilly-sur-Seine
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
- Germany (3):
  - Goethe University Frankfurt, Frankfurt
  - Studiengesellschaft BSF UG (haftungsbeschraenkt), Halle
  - Medizinische Hochschule Hannover, Hanover
- Hungary (4):
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfüred
  - Semmelweis University, Budapest
  - Vasutegeszseguegyi Nonprofit Koezhasznu Kft., Debrecen
  - Győr-Moson-Sopron Vármegyei Petz Aladár Egyetemi Oktató Kórház I. Belgyógyászat, Győr
- Italy (3):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Humanitas Mirasole S.p.A., Rozzano
  - IRCCS Ospedale Sacro Cuore Don Calabria, Verona
- Poland (13):
  - Centrum Medyczne Plejady, Krakow
  - Niepubliczny Zaklad Opieki Zdrowotnej Neuromed M. i M. Nastaj sp. p, Lublin
  - Wojskowy Szpital Kliniczny w Lublinie, Lublin
  - Medicome Sp. z o. o., Oświęcim
  - Trialmed CRS, Piotrkow Trybunalski
  - Termedia Sp. z o.o (NSZOZ Termedica - Centrum Badan Klinicznych), Poznan
  - Ośrodek Badań Klinicznych "METABOLICA", Tarnów
  - Medical Network Sp. z o.o., Warsaw
  - Santa Sp. z o.o., Warsaw
  - Centrum Badan Klinicznych Piotr Napora Lekarze Spolka Partnerska, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
  - LexMedica, Wroclaw
  - Samodzielny PZOZ w Lecznej, Łęczna
- Serbia (2):
  - Kliničko bolnički centar Zvezdara, Belgrade
  - Opšta bolnica "Đorđe Joanović" Zrenjanin Odsek za gastroenterologiju, Zrenjanin
- Slovakia (3):
  - Cliniq s.r.o., Bratislava
  - GASTRO I, s.r.o., Prešov
  - Endomed s.r.o, Vranov nad Topľou
- Slovenia (3):
  - Splošna bolnišnica Celje, Celje
  - Univerzitetni klinični center Maribor, Maribor
  - Splosna Bolnisnica Murska Sobota, Murska Sobota
- Centro Medico Teknon, Barcelona, Spain
- Ukraine (2):
  - Communal non-commercial enterprise "Cherkasy Regional Hospital of Cherkasy regional council", Cherkasy
  - Communal non-commercial enterprise "Khmelnytska Regional Hospital" of Khmelnytskiy regional council, Khmelnytskyi

IPD SHARING:
Plan to Share IPD: No